CLINICAL TRIAL: NCT01705301
Title: Neurotransmitter Measurements Using Wireless Instantaneous Neurotransmitter Concentration System (WINCS) During Deep Brain Stimulation Neurosurgery.
Brief Title: Neurotransmitter Measurements Using (WINCS) During Deep Brain Stimulation Neurosurgery
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Kendall H. Lee, PI, Mayo Clinic
Other Study IDs: 09-007441
Record Dates: First submitted 2012-10-09; First posted 2012-10-12 (Estimated); Last update posted 2017-08-03 (Actual); Status verified 2017-08

CONDITIONS: Essential Tremor; Parkinson's Disease; Dystonia
MeSH Terms: conditions — Essential Tremor; Parkinson Disease; Dystonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Deep Brain Stimulation: Patient's undergoing the clinical procedure of Deep Brain Stimulation will have the experimental protocol that involves, after implantation of the DBS electrodes, a single electrochemical recording electrode, from the WINCS system, implanted along the same trajectory path as the electrophysiology and the DBS electrode
  Interventions: Device: WINCS

INTERVENTIONS:
Device: WINCS — The experimental protocol will involve, after implantation of the DBS electrodes, the patient will have a single electrochemical recording electrode will be implanted along the same trajectory path as the electrophysiology and the DBS electrode

SUMMARY:
In this study, the investigators will monitor extracellular neurotransmitter levels using a probe that is able to perform real time electrochemical detection during deep brain stimulation surgery. The overall question this study is designed to answer is: Are there neurotransmitters released during deep brain stimulation?

DETAILED DESCRIPTION:
In this study, the investigators will monitor extracellular neurotransmitter levels using a probe that is able to perform realtime electrochemical detection during DBS neurosurgery. The overall question this study is designed to answer is: Are there neurotransmitters released during deep brain stimulation? We propose to enroll 45 patients (15 patients each at the three targets for DBS) with Essential Tremor, Parkinson's Disease, and Dystonia who are undergoing DBS neurosurgery. This will be an acute study. Patients with medically identifiable symptoms of the above diseases who have been approved by Mayo DBS committee for implantation of DBS will be selected for this study. These patients will then be consented preoperatively to undergo extracellular electrophysiology which is typical in these cases to determine the target site for implantation of the DBS electrodes. Following this electrophysiologic procedure, the patient will have electrochemical electrode implanted to (1) determine whether there is adenosine release at the site of stimulation during ventral intermediate nucleus (VIM) thalamic DBS, (2) determine whether there is dopamine and adenosine release within the caudate nucleus or putamen during subthalamic nucleus DBS, and (3) determine whether there is dopamine and adenosine release at the site of stimulation during Globus Pallidus DBS.

ELIGIBILITY:
Inclusion Criteria:

* adult Patients with medically intractable Essential Tremor, Parkinson's Disease, and Dystonia who have been approved for DBS surgery by the interdisciplinary Mayo DBS committee.

Exclusion Criteria:

* pregnant patients,
* prisoners,
* children (age less than 18), and
* any patients identified as unsuitable for these protocol by the Mayo DBS committee.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult Patients with medically intractable Essential Tremor, Parkinson's Disease, and Dystonia who have been approved for DBS surgery by the interdisciplinary Mayo DBS committee.
Sampling Method: Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2010-01; Primary Completion 2017-07-27 (Actual); Study Completion 2017-07-27 (Actual)

PRIMARY OUTCOMES:
adenosine release in brain as measured by WINCS (Wireless Instantaneous Neurochemical Concentration Sensing System)recording device | 30 minutes
  Pre, during, post DBS (deep brain stimulation)

SECONDARY OUTCOMES:
dopamine release in brain as measured by WINCS (Wireless Instantaneous Neurochemical Concentration Sensing System)recording device | 30 minutes
  Pre, during, post DBS (deep brain stimulation)

CONTACTS AND LOCATIONS:
Overall Officials: Kendall Lee, MD, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Bennet KE, Tomshine JR, Min HK, Manciu FS, Marsh MP, Paek SB, Settell ML, Nicolai EN, Blaha CD, Kouzani AZ, Chang SY, Lee KH. A Diamond-Based Electrode for Detection of Neurochemicals in the Human Brain. Front Hum Neurosci. 2016 Mar 15;10:102. doi: 10.3389/fnhum.2016.00102. eCollection 2016. PMID 27014033